CLINICAL TRIAL: NCT03861260
Title: To Investigate and Compare The Efficacy of Urethral Dilatation Versus Glycosaminoglycan Layer Replacement in The Management Of Women With Recurrent Urinary Tract Infections
Brief Title: GAG Replacement vs URethral DIlAtatioN
Acronym: GUARDIAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn no participants enrolled
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FAM-99
Record Dates: First submitted 2018-05-03; First posted 2019-03-04 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigid Cystoscopy and Urethral dilatation (Other): Rigid cystoscopy, performed under General Anaesthetic, followed by intervention of urethral dilatation with Hagar dilators.
  Interventions: Procedure: Rigid cystoscopy with urethral dilatation
- Flexible cystoscopy and Glycosaminoglycan Layer replacement (Other): Flexible cystoscopy, under Local Anaesthetic, followed by the intervention, which is 6 installations of Ialuril (a Glycosaminoglycan Layer replacement)
  Interventions: Procedure: Flexible cystoscopy and installation of Glycosaminoglycan layer replacement (laluril)

INTERVENTIONS:
Procedure: Rigid cystoscopy with urethral dilatation — Patients will have a general anaesthetic and a rigid cytoscopic examination of the bladder dilated with sterile water. The urethra will be dilated from FR20 in incremental diameter increases of 2 to French 32 if possible.
  Arms: Rigid Cystoscopy and Urethral dilatation
Procedure: Flexible cystoscopy and installation of Glycosaminoglycan layer replacement (laluril) — Patients will undergo flexible cystoscopy and intravesical installations of Hyaluronic acid (HA) + Chondroitin Sulphate (CS) (GAGs) weekly for 4 weeks and then at 8 weeks and 12 weeks.
  Arms: Flexible cystoscopy and Glycosaminoglycan Layer replacement

SUMMARY:
The aim of this randomised parallel trial is to compare the efficacy of Glycosaminoglycan layer replacement against cystoscopy and urethral dilatation in the treatment of recurrent urinary tract infection in pre-menopausal women.

The women will be randomised to 1 of 2 arms.Arm 1 patients will receive standard treatment from the Urologists. This will involve rigid cystoscopy and urethral dilatation, under general anaesthetic.

Arm 2 patients will receive standard treatment from the Gynaecologists.

DETAILED DESCRIPTION:
Recurrence of a Urinary Tract Infection (UTI) is defined as infection, following complete resolution of a previous UTI.Recurrent UTI (rUTI) is defined as 3 or more microbiologically confirmed UTI within 12 months. rUTI is an economic problem for healthcare services. rUTI is also detrimental to the quality of life (QoL) of women who suffer the disease. 61% of women who suffer rUTI report symptoms of depression and an associated decrease in their reported QoL scores. QoL was found to improve significantly with successful treatment.

E-coli is the most common bacteria causing UTI and 10% are thought to be antibiotic resistant. Consequently, new treatment strategies are required.

The Glycosaminoglycans (GAG) layer is thought to be instrumental as a defence mechanism against uro-pathogens.

GAG's are polysaccharides forming a gel like substance on the apical surface of the bladder wall and act as a barrier to uro-pathogens. There is now strong evidence that a reduction in the impermeability of the GAG layer is linked to rUTI. Urethral dilatation is an alternative treatment to GAG replacement in the management of rUTI. It is a treatment option more widely adopted by Urologists, although there is a paucity of data to support its use.

Currently there is no standardised strategy for the management of women with rUTI. Treatments vary between GAG layer replacement (intravessical therapy with hyaluronic acid and chondroitin sulphate) or a cystoscopy and urethral dilatation. Evidence for each regime varies greatly and is of poor quality. This is a randomised study comparing GAG layer replacement with cystoscopy and urethral dilatation.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Pre-menopausal 3 - 3 episodes of cystitis in the last 12 months as defined by:

   1. 3 symptoms from dysuria, frequency, urgency, suprapubic tenderness, haematuria, polyuria
   2. Or less than 2 symptoms from the above list, but with cloudy urine 4 - Normal flow studies with bladder residual <150ml 5 - Normal renal tract on USS

Exclusion Criteria:

1. - Anatomical anomalies of urinary tract
2. - Neurological condition
3. - Diabetes mellitus
4. - Pregnancy
5. - Use of Immunosuppressants
6. - Symptomatic of UTI at time of treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
The number of Urinary tract infections in the 12 months following treatment | 12 months
  Number of symptomatic UTI episodes in 12 months following treatment

SECONDARY OUTCOMES:
The time to first urinary tract infection after completion of treatment. | 12 month study period
  Time (in days) to first symptomatic UTI episode after completion of treatment.
The change in the Quality of life (QoL) between the time of treatment and at 3, 6 and 12 months following initiation of treatment. | 3, 6 and 12 months
  Following treatment is there any recorded change in the QoL questionnaire (SF-12) score from pre-treatment baseline
The number of adverse events recorded following treatment during the 12-month study period | 12 months
  A record of the number, recorded in groups by their nature, of adverse events following treatment during the 12 month study.
The change in the Patient Satisfaction at 3, 6 and 12 months following initiation of treatment | 3, 6 and 12 months
  Following treatment is there any recorded change in the Patient Satisfaction report from pre-treatment baseline
The change in female sexual function index (FSFI) questionnaire at 3, 6 and 12 months | 3, 6 and 12 months
  Following treatment is there any recorded change in the FSFI questionnaire score (out of 36) from pre-treatment baseline
The change in Hospital anxiety and depression scale (HADS) questionnaire at 3, 6 and 12 months | 3, 6 and 12 months
  Following treatment is there any recorded change in the HADS questionnaire score (out of 21 for anxiety and 21 for depression) from pre-treatment baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Phillips, MBBS MD, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire, United Kingdom